CLINICAL TRIAL: NCT02561104
Title: Outcomes of Resident-Performed Laser-Assisted vs Manual Traditional Phacoemulsification
Brief Title: Resident-Performed Laser-Assisted vs Manual Traditional Phacoemulsification Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 092014-020
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Incipient Cataract; Senile Nuclear Sclerosis
Keywords: cataract; phacoemulsification; laser-assisted surgery; femtosecond laser
MeSH Terms: conditions — Cataract

ARMS (2):
- LenSx (Experimental): Laser-assisted cataract surgery performed using the LenSx femtosecond laser.
  Interventions: Procedure: Laser-assisted cataract surgery.
- Phaco (Experimental): Traditional manual phacoemulsification cataract surgery
  Interventions: Procedure: Traditional manual phacoemulsification

INTERVENTIONS:
Procedure: Laser-assisted cataract surgery.
  Arms: LenSx
Procedure: Traditional manual phacoemulsification
  Arms: Phaco

SUMMARY:
The study design will be a prospective study comparing laser-assisted cataract extraction cases and traditional manual phacoemulsification cases. All cases will be performed by faculty-supervised residents at Parkland Memorial Hospital. This study aims to examine visual acuity and complication rates in femtosecond laser-assisted cataract surgery compared to traditional manual phacoemulsification cataract surgery for the beginning surgeon. In addition, this study will assess the subjective novice surgeon experience and the patient experience in terms of expectations and results.

DETAILED DESCRIPTION:
The study design will be a prospective study comparing laser-assisted cataract extraction cases and traditional manual phacoemulsification cases. All cases will be performed by faculty-supervised residents at Parkland Memorial Hospital. Cataract surgery training is a standard requirement of all ophthalmology residents who are part of this clinical study.

Each resident must be a post graduate year 4 (PGY-4) level resident before being asked to be a part of this clinical study. Typically, each resident will have completed approximately 30 cataract surgeries by their PGY-3 residency year of training. These traditional phacoemulsification require manual capsulorrhexis creation with which residents will have experience prior to study participation. Other critical manual surgical steps of traditional and femtosecond-laser assisted cataract surgery require similar surgical skill sets, thus residents should have surgical skills applicable to both techniques prior to study involvement.

In addition to performing 30 traditional phacoemulsification surgeries, residents also will have assisted with femtosecond laser-assisted cases during their PGY-3 training year training at the Dallas VA medical center and with staff at University of Texas (UT) Southwestern Medical Center during their cornea rotation. The femtosecond-assisted cases completed by each resident in the study at Parkland will be the Alcon Certification cases for each resident. Performing femtosecond-laser assisted cases at this level of training will provide objective insights into this new surgical technique in resident hands. Patients will not be subjected to any additional risk due to participation in this study as femtosecond laser Alcon Certification is already being performed by residents as part of their standard UT Southwestern ophthalmology training.

Patient eyes that meet the inclusion and exclusion criteria below will be randomly assigned to either the laser-assisted or the standard manual phacoemulsification group based. Following surgery, patients will return for post-operative visits at post-op day 1, post-op week 1, post-op month 1, and post-op month 3. Subjects will be followed in the Parkland Surgery Chief clinic. Subjects will not necessarily see the same study surgeon during each post-operative visit period. It should be noted this is the standard procedure as currently practiced in the Parkland ophthalmology clinic.

Verification of subject adherence to the post-operative follow-up visit schedule will be overseen by the PI throughout the course of the project. Weekly communication with sub-investigators will take place in order to review any outstanding concerns including recruitment effort, surgery schedules, and post-operative visit timelines. Arrangements for additional visits will also be reviewed and scheduled if medically necessary depending on individual patients' post-operative clinical course. Patients will be assigned to each group during the period of September 2015 through July 2016 and followed as part of the study for 3 months post-operatively.

Patients will be offered the same kerato-refractive procedures including manual limbal relaxing incisions or LenSx astigmatic keratotomy that would be offered to patients who are not part of this study. Patients will also be evaluated for benefit from advanced technology intraocular lenses (Toric for astigmatism and ReStor multifocal) that patients who are not part of the study would be offered. Offering advanced technology lenses or combined kerato-refractive procedures is not expected to influence the visual acuity study outcomes for patients in this study. Patient's clinical history, past medical history and ophthalmic medical notes (in particular pre-operative evaluation, operative, and post-operative follow up) will be reviewed. De-identified data points will be extracted for this project.

ELIGIBILITY:
Inclusion Criteria:

1. Referred for cataract surgery at Parkland Memorial Hospital
2. Potential post-operative visual acuity of 20/30 or greater determined by potential acuity meter (PAM) testing or modified super pinhole potential acuity of 20/30 or greater
3. Clear intraocular media other than cataract in study eye(s)
4. Subject eyes will have a dilated pupil diameter of at least 6 mm
5. Subject eyes will lack other pre-existing ocular pathology or condition that may confound treatment effects, including diabetic retinopathy, previous retinal detachment, iris neovascularization, amblyopia, optic nerve atrophy or recurrent severe anterior or posterior segment inflammation of unknown etiology.

Exclusion Criteria:

1. Severe corneal diseases or prior corneal surgery
2. Active, significant external ocular or eyelid disease
3. History of lens abnormalities including posterior polar cataract and zonular weakness precluding standard non-complex cataract surgery
4. Retinal or posterior segment disease
5. Advanced glaucoma, white or advanced cataract (precluding adequate examination of the posterior pole)
6. Anatomic conditions that prevent placement of the femtosecond laser docking ring
7. Corneal opacity that will interfere with the laser beam (hazy cornea)
8. Presence of blood or materials in the anterior chamber
9. Hypotony, advanced glaucoma, or presence of cornea implant
10. Poor dilating pupil such that the iris is not peripheral to the intended diameter for the capsulotomy
11. Condition which would cause inadequate clearance between the intended capsulotomy depth and the corneal endothelium
12. Any contraindication to cataract or kerato-refractive surgery
13. Contact lens wearers must discontinue the use of contacts for an appropriate period of time to ensure that their corneas are stable before screening measurements are performed. For rigid gas permeable (RGP) lenses, it is at least 2-4 weeks before accurate imaging measurements can be performed. Study doctor will assess patient findings and determine how long RGP lens wear must be discontinued prior to surgery. For soft contact lenses, it is at least 3 days prior to study measurements.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Complication rates | Operative visit to last post-op visit at 3 mos
  Complication and adverse event monitoring will occur at each visit: pre-operative, operative, post-op day 1, post-op day 7-14, post-op day 30-60 and 3 mos post-op
Visual Acuity | Change between baseline and 3 mos post-op.
  Bilateral best spectacle corrected visual acuity

SECONDARY OUTCOMES:
Patient benefit perception | Post-op day 1
  Patient perception of results assessed by questionnaire
Patient benefit perception | Post-op day 30-60
  Patient perception of results assessed by questionnaire
Patient benefit perception | 3 mos post-op
  Patient perception of results assessed by questionnaire
Corneal Endothelial Cell Count (ECC) | Change from baseline to post-op day 30-60
  Specular micrography performed at baseline and post-op day 30-60 OR 3 month post-op* to measure change in ECC
  *3 month ECC test will be done only if test was unable to be performed on post-op day 30-60 visit
Lens removal time | Operative visit
  Comparison of time required for nuclear and cortex removal using the two techniques

CONTACTS AND LOCATIONS:
Overall Officials: Brock Hansen, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States